CLINICAL TRIAL: NCT01948011
Title: Study of the Racecadotril Linearity After Single Administrations of 10, 30 and 60 mg of a New Racecadotril Formulation (Suspension) by Oral Route and Evaluation of the Comparative Bioavailability of This New Formulation Versus the Sachet Formulation (Granules) After a 60 mg Single Oral Administration in Healthy Male Volunteers
Brief Title: Racecadotril Suspension Linearity Study & Comparative Bioavailability Versus Granules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: P13-01 / BP0.52; 2013-002746-36 (EudraCT Number)
Record Dates: First submitted 2013-09-11; First posted 2013-09-23 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Male Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Racecadotril 10mg suspension (Experimental): single oral dose
  Interventions: Drug: Racecadotril granules
- Racecadotril 30mg suspension (Experimental): single oral dose
  Interventions: Drug: Racecadotril granules
- Racecadotril 60mg suspension (Experimental): single oral dose
  Interventions: Drug: Racecadotril granules
- Racecadotril 60mg granules (Active Comparator): single oral dose
  Interventions: Drug: Racecadotril suspension

INTERVENTIONS:
Drug: Racecadotril suspension — Racecadotril suspension at 10, 30 and 60mg. Single oral dose.
  Arms: Racecadotril 60mg granules
Drug: Racecadotril granules — Racecadotril granules at 60mg. Single oral dose.
  Arms: Racecadotril 10mg suspension; Racecadotril 30mg suspension; Racecadotril 60mg suspension

SUMMARY:
To investigate the Racecadotril pharmacokinetic linearity after single oral administration of 10, 30 and 60 mg as a suspension.

To evaluate the comparative bioavailability of the new Racecadotril formulation (suspension) versus the reference sachet formulation (granules)

DETAILED DESCRIPTION:
This is a single center, open-label, single oral dose, 4-period cross-over study to assess the bioequivalence of a new formulation (suspension) in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male,
* 18 to 45 years old,
* be certified as normal by a comprehensive clinical assessment (detailed medical history and a complete physical examination), arterial blood pressure (BP), heart rate (HR), an ECG and laboratory investigations (haematological, blood chemistry tests, urinalysis), the results of which are within the normal range and/ or judged by the investigator as clinically acceptable for healthy subjects,
* Body Mass Index (BMI) between 18 and 28 kg/m2.

Exclusion Criteria:

* History of cardiovascular, pulmonary gastro-intestinal, hepatic, renal, metabolic, haematological, neurological, psychiatric, systemic, or infectious disease.
* Any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Subject has used any drug including OTC products two weeks before the scheduled administration of study drug, except paracetamol (maximum 1g/day).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Bio-equivalence | Total study duration per subject should be 6 weeks.
  Several blood sample will be collected at each period to investigate the racecadotril pharmacokinetic linearity and to evaluate the comparative bioavalibility.
  4-period, cross over, single oral dose at each period.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, MD, Principal Investigator — Eurofins Optimed
Locations (1):
- Eurofins Optimed, Gières, France